CLINICAL TRIAL: NCT03349619
Title: ReNIM Study - Nebulized Resveratrol Plus Carboxymethyl-β-Glucan for Reducing Nasal Interleukin-5 (IL-5) Measurements in Children With Allergic Rhinitis
Brief Title: Nebulized Resveratrol Plus Carboxymethyl-β-Glucan for Reducing IL-5 in Children With Allergic Rhinitis
Acronym: RENIM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Ph.D. Senior Researcher. Coordinator of Pediatric Allergy and Asthma Research Group. Institute of Biomedicine and Molecular Immunology, IBIM, National Research Council of Palermo, Italy., Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10/2017
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol plus Carboxymethyl-β-Glucan (Experimental)
  Interventions: Drug: Resveratrol plus Carboxymethyl-β-Glucan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resveratrol plus Carboxymethyl-β-Glucan — Patients in this arm will receive Resveratrol plus Carboxymethyl-β-Glucan, two sprays (100µL/spray) per nostril three times/day for 4 weeks
  Arms: Resveratrol plus Carboxymethyl-β-Glucan
Drug: Placebo — Patients in this arm will receive nasal saline solution 0.9%, two sprays per nostril, three times/day for 4 weeks
  Arms: Placebo

SUMMARY:
Single-center, randomized, placebo-controlled study to:

* characterize the subjects at baseline and discriminate groups of children based on IL-5, IL-17, IL-23 and INF-γ;
* investigate the effect of Resveratrol plus Carboxymethyl-β-Glucan, two sprays (100µL/spray) for nostril three times/day for 4 weeks, in comparison with placebo, in reducing nasal interleukin-5 (IL-5) in children with Allergic Rhinitis (AR).

Secondary objectives are to examine the effect of resveratrol plus carboxymethyl-β-glucan, in comparison with placebo, on subjective parameters, i.e. symptom scores, visual analogue scales for rhinitis, quality of life and quality of sleep, and the effect on objective parameters, i.e. nasal nitric oxide (nNO) levels, nasal cytology and acoustic rhinometry.

ELIGIBILITY:
Inclusion Criteria:

* history of AR in the previous year;
* positive skin prick test to seasonal allergens.

Exclusion Criteria:

* acute upper respiratory infections in the last 4 weeks;
* lifetime history of asthma (doctor diagnosis);
* use of nasal or oral corticosteroids, nasal or oral decongestants, antihistamines in the last 4 weeks;
* anatomic nasal defects (ie, septum deviation), or nasal polyps;
* active smoker.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Nasal Interleukin-17 (IL-17) | Baseline
  IL-17 level at baseline
Nasal Interleukin-23 (IL-23) | Baseline
  IL-23 level at baseline
Nasal Interferon-γ (INF-γ) | Baseline
  INF-γ level at baseline
Nasal PH | Baseline
  Nasal PH at baseline
Nasal Interleukin-5 (IL-5) | Baseline and 28 days
  Mean change in IL-5 level from baseline to the end of treatment.

SECONDARY OUTCOMES:
Total 5 Symptom Score (T5SS) | Baseline and 28 days
  Mean change in T5SS score from baseline to the end of treatment.
Visual Analogue Scale for Rhinitis (VAS) | Baseline and 28 days
  Mean change in VAS score from baseline to the end of treatment.
Paediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) | Baseline and 28 days
  Mean change in PRQLQ score from baseline to the end of treatment.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 28 days
  Mean change in PSQI score from baseline to the end of treatment.
Nasal Exhaled Nitric Oxide (nNO) | Baseline and 28 days
  Mean change of nNO from baseline to the end of treatment.
Nasal Cytology | Baseline and 28 days
  Mean change in nasal cytology counts from baseline to the end of treatment.
Acoustic Rhinometry: Minimal Cross-sectional Area (MCA) | Baseline and 28 days
  Mean change of MCA from baseline to the end of treatment.
Acoustic Rhinometry: Nasal Volume from the first 5 cm from the nostril (V.0-5) | Baseline and 28 days
  Mean change of V.0-5 from baseline to the end of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Biomedicine and Molecular Immunology (IBIM) - National Research Council of Palermo, Palermo, Italy